CLINICAL TRIAL: NCT06191692
Title: An Open-label, Randomized Controlled Trial of the New One-month Regimen Versus the Current Three-month Regimen for the Treatment of Tuberculosis Infection in Vietnam
Brief Title: 1HP Versus 3HR in the Treatment of Tuberculosis Infection in Vietnam
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Freundeskreis Für Internationale Tuberkulosehilfe e.V (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBIshort
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis Infection
Keywords: Tuberculosis; TB preventive therapy; Tuberculosis infection; Latent TB infection; LTBI; TBI
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid; rifapentine; Rifampin

STUDY DESIGN:
Intervention Model Description: Households will be randomized in a 1:1 ratio to the two treatment groups (1HP/3HR) using cluster randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months of daily rifampicin plus isoniazid regimen (Arm A) (Active Comparator): Participants will receive rifampicin (dosage based on their weight*, 10mg/kg/day, maximum 600mg), 300 mg of isoniazid, and 25 mg or 50 mg of pyridoxine (vitamin B6) each day from week 1 to week 12 for a total of 90 doses.
  * Weight will be monitored and dosing adjusted as needed during treatment
  Interventions: Drug: Isoniazid; Drug: Rifampicin
- 1 month of daily rifapentine plus isoniazid regimen (Arm B) (Experimental): Participants will receive rifapentine (dosage based on their weight* 300 mg daily for participants body weight of 30kg -<35 kg, 450 mg daily for a weight of 35 to 45 kg, and 600 mg for a weight of >=45 kg), 300 mg of isoniazid, and 25 mg or 50 mg of pyridoxine (vitamin B6) each day from week 1 to week 4 for a total of 28 days.
  * Weight will be monitored and dosing adjusted as needed during treatment
  Interventions: Drug: Isoniazid; Drug: Rifapentine

INTERVENTIONS:
Drug: Isoniazid — This randomized control trial will compare the treatment adherence and safety of the 1HP (Arm B) regimen and standard 3HR (Arm A) regimens for TB infection treatment
  Other Names: INH
Drug: Rifapentine — This randomized control trial will compare the treatment adherence and safety of the 1HP (Arm B) regimen and standard 3HR (Arm A) regimens for TB infection treatment
  Other Names: RPT
  Arms: 1 month of daily rifapentine plus isoniazid regimen (Arm B)
Drug: Rifampicin — This randomized control trial will compare the treatment adherence and safety of the 1HP (Arm B) regimen and standard 3HR (Arm A) regimens for TB infection treatment
  Other Names: RIF
  Arms: 3 months of daily rifampicin plus isoniazid regimen (Arm A)

SUMMARY:
Introduction: Tuberculosis (TB) infection is a key driver of the TB pandemic, with over 10.6 million people fell ill with TB disease in 2022. About one-quarter of the global population is estimated to be infected with TB bacteria. Around 5-10% of people with TB infection will develop active and contagious TB disease, which could be largely avoided if TB infection is identified and given effective preventative treatment, before progression to active disease. The long treatment of TB infection with regimens lasting from three to nine months is a significant barrier to treatment completion in individuals with a confirmed diagnosis of TB infection. Adapting a shorter regimen than the current regimens could lead to a higher treatment completion rate and increased uptake of preventative therapy for TB, as well as reduced side effects.

Methods and analysis: An open-label, randomized clinical trial (1:1) will be performed in two study sites in Ha Noi, Vietnam (Vietnam National Lung Hospital and Ha Noi Lung Hospital). Adult household contacts (n=350) of people with new, bacteriologically-confirmed, pulmonary, drug-susceptible TB who initiate treatment will be invited to participate.

Aim: To compare the TB preventive therapy completion rates and adverse event incidence between a new one-month regimen (1HP) versus the current three-month regimen (3HR)*.

*1HP= one month of daily isoniazid (H/INH) and rifapentine (P/RPT) 3HR= three months of daily isoniazid (H/INH) and rifampicin (R/RIF)

DETAILED DESCRIPTION:
Latent TB infection, hereafter referred to as TB infection, is a key driver of the TB pandemic. Over 10.6 million people developed active TB in 2022 and about one-quarter of the global population is estimated to be infected with TB bacteria, meaning approximately two billion people are affected worldwide. On average, 5-10% of people with TB infection will develop active TB, usually within the first five years after their initial TB infection. Therefore, preventative treatment is a fundamental component of a comprehensive strategy to end TB.

The current duration of TB Prevention Treatment (TPT), which lasts from three to nine months, is a significant barrier resulting in the low uptake of the TPT.

A one-month TPT regimen using two drugs (isoniazid and rifapentine, 1HP) was proven effective and had higher completion rates for people living with HIV; however, the initial demonstration trial was not performed in a cohort of people without HIV. The use of a shorter TPT regimen than the current three-month TPT regimen could lead to higher completion rates and increased uptake among a large number of individuals in need of TPT. Moreover, it may potentially reduce adverse events as well as decrease the medical and non-medical costs associated with the TPT.

Therefore, the investigators propose a comprehensive study of shortened TPT for TB infection in Vietnam, a low HIV burden setting.

An open-label, randomized controlled trial (TBIshort) of the new one-month TPT regimen versus the current three-month regimen for the treatment of TB infection in Vietnam will be performed and funded by Stop TB Partnership's TB REACH initiative to compare treatment completion rate and safety between the two regimens. Households will be randomized in a 1:1 ratio to the two arms using cluster randomization. All participants from the same household will be allocated to the same treatment regimen arm. The proposed study will address key knowledge gaps, and provide objective evidence to guide decision-making for the use of the 1HP regimen for the treatment of TB infection in a low HIV burden setting.

Aims

1. Main objective:

   Objective 1: Compare the treatment adherence and safety of the 1HP regimen and the standard 3HR regimen for TB infection treatment
2. Specific objectives:

Objective 2: Compare the treatment completion rates for TB infection between 1HP and 3HR regimens.

Objective 3: Compare adverse events incidence for 1HP and 3HR regimens during three months from treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Household contacts of people with new, bacteriologically-confirmed, pulmonary, drug-susceptible TB who initiated treatment with residence in the intervention areas;
* Positive QFT-Plus or TST results (TST induration of at least 5mm)
* Agree to remain in contact and provide updated information as necessary, and have no current plans to relocate outside the designed area for the duration of the study;
* Age ≥ 18 years;
* Capable of providing signed informed consent;
* Willing to participate in the study visits and procedures

Exclusion Criteria:

* Indeterminate results on QFT-Plus;
* Clinical or radiographic suspicions or history of previous active TB;
* Known hypersensitivity or contraindication to any components of the regimens;
* Weight <30kg;
* Acute or chronic liver failure with elevated liver enzymes or evidence of liver dysfunction such as jaundice or a history of liver failure caused by isoniazid or rifampicin; History of liver cirrhosis at any time before study entry;
* Infection with suspected or confirmed tuberculosis strains resistant to isoniazid or rifampicin;
* Porphyria- Porphyrin metabolism disorder;
* Polyneuropathy (self-reported/ confirmed);
* Pregnant or planning to become pregnant within 120 days of enrollment;
* Any other severe underlying condition that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial;
* Participation in other clinical intervention trials or research protocols (participation in other studies that do not involve an intervention may be allowed, but this must be discussed and approved by the Chief Investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
1. % Adequate adherence in each arm | From study entry at Week 0 through up to 16 weeks of 3HR (Arm A), or up to 6 weeks of 1HP (Arm B), to be reported at the end of the trial.
  Adequate treatment adherence is defined as taking ≥90% of TB preventive therapy doses within the time frame. Treatment adherence will be recorded by both study schedule and programmatic adherence.

SECONDARY OUTCOMES:
The incidence rate of severe adverse events among two arms. | From study entry at Week 0 through up to 16 weeks of 3HR (Arm A), or up to 6 weeks of 1HP (Arm B)
  Severe adverse events are defined (DAIDS) as any untoward medical occurrence that, at any dose:
  * Results in death
  * Life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Congenital anomaly/birth defect
Comparison of adherence measured as the proportion of treatment taken in the regimens (1HP vs 3HR). | From study entry at Week 0 through up to 16 weeks of 3HR (Arm A), or up to 6 weeks of 1HP (Arm B)
The incidence rate of a targeted event of grade 3,4 or 5*** and one grade increase from the baseline among two arms. | From study entry at Week 0 through up to 16 weeks of 3HR (Arm A), or up to 6 weeks of 1HP (Arm B)
  Targeted event includes:
  1. Flu-like symptoms including weakness, fatigue, nausea, vomiting, headache, fever, aches, sweats, dizziness, shortness of breath, flushing, or chills.
  2. Hepatotoxicity, defined as a five-fold or greater increase in the AST/ALT level, a three-fold or greater increase with clinical symptoms, or total bilirubin level > 51.3 micromole/L.
  3. Peripheral neuropathy (Clinical diagnosis)

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Vietnam National Lung Hospital, Hanoi, Hanoi
  - Ha Noi Lung Hospital, Hà Nội

IPD SHARING:
Plan to Share IPD: No